CLINICAL TRIAL: NCT02557139
Title: A 3-way, Crossover, Randomized, Open-label Study in Healthy Subjects Comparing the Bioavailability of Belumosudil (KD025) Tablets in Fed and Fasted States and Relative Bioavailability of Tablets and Capsules in the Fed State
Brief Title: Bioavailability of Belumosudil (KD025) in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KD025-106; 2015-002832-42 (EudraCT Number)
Record Dates: First submitted 2015-09-01; First posted 2015-09-23 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Bioavailability
MeSH Terms: interventions — belumosudil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regimen A (Experimental): Single-dose belumosudil 200 mg tablet in the fasted state
  Interventions: Drug: Belumosudil Tablet
- Regimen B (Experimental): Single-dose belumosudil 200 mg tablet in the fed state
  Interventions: Drug: Belumosudil Tablet
- Regimen C (Experimental): Single-dose belumosudil capsules (administered as two 100-mg capsules) in the fed state
  Interventions: Drug: Belumosudil Capsule

INTERVENTIONS:
Drug: Belumosudil Tablet
  Other Names: Rezurock (brand); SLx-2119
  Arms: Regimen A; Regimen B
Drug: Belumosudil Capsule
  Other Names: Rezurock (brand); SLx-2119
  Arms: Regimen C

SUMMARY:
Phase 1 bioavailability study to evaluate the pharmacokinetics (PK) and tolerability/safety of the belumosudil tablet formulation in the fasted and fed states and compared to the belumosudil capsule formulation in the fed state.

DETAILED DESCRIPTION:
This is a Phase 1, 3-way, crossover, randomized, open-label study in healthy subjects designed to compare the bioavailability of belumosudil (previously known as KD025) tablet formulation administered in the fed and fasted states and to assess the relative bioavailability of belumosudil tablet and capsule formulations in the fed state.

The primary objective of the study is to determine the PK parameters of belumosudil tablet formulation in the fed and fasted states.

The secondary objectives of the study are: (1) to assess the relative bioavailability of a tablet (test) to capsule (reference formulation of belumosudil; (2) to assess and compare the variability in the maximum concentration (Cmax) and area under the concentration-time curve (AUC) for belumosudil treatments (belumosudil 200 mg tablet in the fasting state, belumosudil 200 mg tablet in the fed state, and belumosudil as two 100 mg capsules in the fed state); and (3) to provide additional safety and tolerability information for belumosudil.

This is a single-center, open-label, randomized, single-dose, 3-period, 3-way, crossover study in healthy subjects.

In each of 3 study periods, each subject receives 1 of the following single-dose treatments:

* Regimen A: Belumosudil 200 mg tablet in the fasted state
* Regimen B: Belumosudil 200 mg tablet in the fed state
* Regimen C: Belumosudil 200 mg as two 100-mg capsules in the fed state

Subjects are randomized to receive 1 dose of investigational product (IP; belumosudil tablet or capsule) in the morning of Day 1 in a randomized manner following an overnight fast or a high-fat breakfast. Administration is performed on Day 1 with an appropriate interval between subjects based on logistical requirements. Start time is determined based on logistics.

Subjects undergo a screening visit in the 21 days preceding first dose. Subjects are admitted to the clinical unit on the evening prior to dosing (Day -1), remain on site until 24 hours post-dose, and return to the clinic at 36 and 48 hours post-dose for PK assessments.

There is a minimum washout period of 6 days between each dose administration. All other meals are standardized for each of the in-clinic phases of the 3 treatment periods. Each period follows the same study design.

The randomized cohorts for the 3-periods were as follows:

* Cohort ABC: Regimen A (Period 1); Regimen B (Period 2); Regimen C (Period 3)
* Cohort BCA: Regimen B (Period 1); Regimen C (Period 2); Regimen A (Period 3)
* Cohort CAB: Regimen C (Period 1); Regimen A (Period 2); Regimen B (Period 3)

A follow-up call is made 3 to 5 days after the final dose of IP.

Planned enrollment is 24 subjects to insure there are 20 evaluable subjects. A subject is considered evaluable if (s)he completes treatment with fasted and fed tablet formulations (Regimens A and B) without major protocol deviations.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study entry subjects has to satisfy all of the following criteria:

1. Healthy males
2. Aged 18 to 55 years of age
3. Good state of health (mentally and physically) as indicated by a comprehensive clinical assessment (detailed medical history and a complete physical examination), ECG, and laboratory investigations (hematology, coagulation, clinical chemistry and urinalysis)
4. Body mass index 18.0-30.0 kg/m^2, or if outside the range, considered not clinically significant by the Investigator
5. Willing and able to communicate and participate in the whole study
6. Provide written informed consent
7. Agree to use an adequate method of contraception for up to 90 days post discharge

Exclusion Criteria

Subjects are excluded from the study if one of more of the following statements is applicable:

1. Participated in a clinical research study within the previous 3 months
2. Study site employees, or immediate family members of a study site or sponsor employee
3. Had been previously enrolled in this study
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption > 21 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
6. Current smokers and those who had smoked within the last 12 months. A breath carbon monoxide (CO) reading of greater than 10 ppm at screening
7. Did not have suitable veins for multiple venepunctures/cannulation as assessed by the Investigator at screening
8. Clinically significant abnormal biochemistry, hematology, coagulation, or urinalysis as judged by the Investigator
9. Positive drugs of abuse test result or alcohol breath test
10. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody (Ab) or human immunodeficiency virus (HIV) results
11. History of any clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal (GI) disease that may have compromised the subject's safety or interfered with the objectives of the study as judged by the investigator
12. Subject had a history or presence of any of the following:

    * Active GI disease requiring therapy
    * Hepatic disease and/or alanine aminotransaminase (ALT) or aspartate aminotransaminase (AST) > 1.5 × upper limit of normal (ULN) at screening
    * Renal disease and/or serum creatinine > 1.5 × ULN at screening
    * Other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs
13. QT interval corrected using Fridericia's formula (QTcF) > 450 msec at the screening or admission ECG
14. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
15. Known sensitivity to ROCK2 inhibitor agents or to any of the constituents of the belumosudil formulation
16. Presence or history of clinically significant allergy requiring treatment, as judged by the Investigator. Hayfever is permitted unless it is active.
17. Donation or loss of > 400 mL of blood within the previous 3 months
18. Taking or had taken any prescribed or over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies in the 14 days before IP administration
19. Fails to satisfy the Investigator's discretion of fitness to participate or for any other reason

Additional Restrictions

1. Abstain from alcohol during the 24 h prior to each admission until discharge from the clinic in each study period
2. Not to drink liquids or eat food containing grapefruit, cranberry, caffeine, or other xanthines from 24 hours prior to each admission until 48 hours post-dose
3. Refrain from eating food containing any seeds (e.g., poppy) for 48 hours before the screening visit and then from 48 h prior to each admission until discharge from the clinic for each study period
4. Not to take part in any unaccustomed strenuous exercise from 72 hours prior to the screening visit and then from 72 hours prior to admission until discharge from the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10-12 (Actual); Study Completion 2015-10-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical Limited, Ruddington Nottingham, United Kingdom

REFERENCES:
- [Background] Schueller O, McDermott J, Evans P, Lohmer L, Alabanza A, Patel J. Phase 1 Studies to Evaluate the Food Effect and Relative Bioavailability of Tablet and Capsule Formulations of Belumosudil in Healthy Adult Subjects. Clin Pharmacol Drug Dev. 2022 Jul;11(7):807-814. doi: 10.1002/cpdd.1083. Epub 2022 Mar 2. PMID 35238174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment: 23 subjects
Groups:
- Cohort ABC: Period 1: Single-dose Belumosudil 200 mg tablet fasted (Regimen A); Washout; Period 2: Single-dose Belumosudil 200 mg tablet fed (Regimen B); Washout; Period 3: Single-dose Belumosudil two 100-mg capsules, i.e., 200 mg (Regimen C)
- Cohort BCA: Period 1: Belumosudil 200 mg tablet fed; Washout; Period 2: Belumosudil 200 mg by capsule, i.e., two 100-mg capsules fed; Washout; Period 3: Belumosudil 200 mg tablet fasted
- Cohort CAB: Period 1: Single-dose Belumosudil 200 mg by capsule, i.e., two 100-mg capsules fed; Washout; Period 2: Single-dose Belumosudil 200 mg tablet fasted; Washout; Period 3: Single-dose Belumosudil 200 mg tablet fed
Period: Overall Study
Arm/Group | Cohort ABC | Cohort BCA | Cohort CAB
Started | 8 | 8 | 7
Completed | 6 | 8 | 5
Not Completed | 2 | 0 | 2
Not completed — Significant liver elevation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Illness of prohibited medication | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort ABC | Cohort BCA | Cohort CAB | Total
Number analyzed (Participants) | 8 | 8 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.1 (11.0) | 32.3 (12.4) | 43.0 (9.0) | 36.2 (11.5)
Age, Continuous [Median (Full Range); unit: Years] | 32.5 [20 to 53] | 27.5 [21 to 50] | 46.0 [30 to 54] | 33.0 [20 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 8 | 7 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 7 | 7 | 6 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI (body mass index) [Mean (Standard Deviation); unit: kg/m^2] | 26.19 (2.67) | 25.79 (2.43) | 26.53 (3.35) | 26.15 (2.70)
BMI (body mass index) [Median (Full Range); unit: kg/m^2] | 26.4 [22.4 to 29.3] | 26.0 [22.6 to 28.7] | 26.1 [22.1 to 30.0] | 26.10 [22.1 to 30.0]

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Cmax of Dosing Regimen A (Tablets--Fasting) vs. Dosing Regimen B (Tablets--Fed) for KD025, KD025m1, and KD025m2 at 48 Hours Post-dose
Description: Maximum concentration (Cmax) of parent drug (KD025), Metabolite 1 (KD025m1), and Metabolite 2 (KD025m2) when administering a single dose of belumosudil 200 mg tablet to subjects who are fasting (Regimen A) compared to administering a single dose of belumosudil 200 mg tablet to subjects who are fed (Regimen B) at 48 hours after dosing
Time Frame: Pre-dose (0), and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours post-dose
Population: Not all subjects received each regimen.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Regimen A: Single-dose belumosudil 200 mg tablet in the fasting state
- Regimen B: Single-dose belumosudil 200 mg tablet in the fed state
  Belumosudil Tablet
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 23 | 20
ng/mL
  Cmax: KD025 | 821 (129.5) | 2100 (49.8)
  Cmax: KD025m1: number analyzed (Participants) | 16 | 20
  Cmax: KD025m1 | 19.4 (51.6) | 25.8 (42.0)
  Cmax: KD025m2: number analyzed (Participants) | 22 | 20
  Cmax: KD025m2 | 173 (122.6) | 412 (63.0)

2. Primary Outcome: Pharmacokinetics: AUCs of Dosing Regimen A (Tablets--Fasting) vs. Dosing Regimen B (Tablets--Fed) for KD025, KD025m1, and KD025m2 at 48 Hours Post-dose
Description: Area under concentration-time curve from zero to last dose of belumosudil 200 mg tablets (AUC[0-last]) and from zero to infinity (AUC[0-inf]) for Metabolite 1 (KD025m1), and Metabolite 2 (KD025m2) when administering a single dose of belumosudil 200 mg tablet to subjects who are fasting (Regimen A) compared to administering a single dose of belumosudil 200 mg tablet to subjects who are fed (Regimen B) at 48 hours after dosing
Time Frame: Pre-dose (0), and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours post-dose
Population: Not all subjects in either cohort had all AUC measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h)/mL
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 23 | 20
(ng*h)/mL
  AUC(0-last): KD025 | 4520 (121.3) | 9750 (49.3)
  AUC(0-last): KD025m1: number analyzed (Participants) | 16 | 20
  AUC(0-last): KD025m1 | 19.8 (150.6) | 45.2 (95.3)
  AUC(0-last): KD025m2: number analyzed (Participants) | 22 | 20
  AUC(0-last): KD025m2 | 550 (133.3) | 1320 (62.6)
  AUC(0-inf): KD025: number analyzed (Participants) | 14 | 17
  AUC(0-inf): KD025 | 4910 (146.9) | 10100 (52.9)
  AUC(0-inf): KD025m1: number analyzed (Participants) | 1 | 1
  AUC(0-inf): KD025m1 | 153 (0) | 98.7 (0)
  AUC(0-inf): KD025m2: number analyzed (Participants) | 16 | 17
  AUC(0-inf): KD025m2 | 691 (76.7) | 1370 (62.6)

3. Secondary Outcome: Pharmacokinetics: Cmax for the Relative Bioavailability of Regimen B/Regimen A and Regimen B/Regimen C by Ratio of the Adjusted Geometric Means at 48 Hours Post-dose
Description: Analysis of the maximum concentration (Cmax) of the relative bioavailability of Regimen B (belumosudil 200 mg tablet-fed) vs. Regimen A (belumosudil 200 mg tablet-fasting) and for Regimen B vs. Regimen C (belumosudil 200 mg capsule-fed) utilizing the Ratio of the Adjusted Geometric Means at 48 hours after dosing
Time Frame: Pre-dose (0), and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours post-dose
Measure: Number (90% Confidence Interval); unit: Ratio of Adjusted Geometric Means
Groups:
- Regimen B/Regimen A: Single-dose belumosudil 200 mg tablet fed (Regimen B) divided by single-dose belumosudil 200 mg tablet fasting (Regimen A)
- Regimen B/Regimen C: Single-dose belumosudil 200 mg tablet fed (Regimen B) divided by single-dose belumosudil 200 mg capsule fed (Regimen C)
Arm/Group | Regimen B/Regimen A | Regimen B/Regimen C
Number analyzed (Participants) | 20 | 20
Ratio of Adjusted Geometric Means | 225.02 [176.08 to 287.57] | 119.38 [93.41 to 152.56]
Statistical Analysis 1: Comparison: Regimen B/Regimen A; Cmax null hypothesis: Ratio of Adjusted Geometric Means = 100%; Test type: Equivalence — If the 90% confidence interval for the comparison of fed vs. fasted is within the acceptance range 80.00% to 125.00%, then it is concluded that there is no effect of food on belumosudil tablets; p < 0.001, t-test, 2 sided; Ratio of Adjusted Geometric Means (%) = 100, 90% CI 2-sided [80.00 to 125.00]; Intra-subject variability: 48.00%
Statistical Analysis 2: Comparison: Regimen B/Regimen C; Cmax null hypothesis: Ratio of Adjusted Geometric Means = 100%; Test type: Equivalence — If the 90% confidence interval for the comparison of belumosudil tablet (test drug) vs. the belumosudil capsule (reference drug) is within the acceptance range 80.00% to 125.00%, then it is concluded that there is no effect on the use of belumosudi tablet compared to belumosudil capsule; p = 0.23, t-test, 2 sided; Ratio of Geometric Means (%) = 100, 90% CI 2-sided [80.00 to 125.00]; Intra-subject variability: 48.00%

4. Secondary Outcome: Pharmacokinetics: AUCs for the Relative Bioavailability of Regimen B/Regimen A and Regimen B/Regimen C by Ratio of the Adjusted Geometric Means at 48 Hours Post-dose
Description: Analysis of the area under concentration-time curve for zero to infinity (AUC[0-inf]), and zero to last dose (AUC[0-last]) of the relative bioavailability of Regimen B (belumosudil 200 mg tablet-fed) vs. Regimen A (belumosudil 200 mg tablet-fasting) and for Regimen B vs. Regimen C (belumosudil 200 mg capsule-fed) utilizing the Ratio of the Adjusted Geometric Means at 48 hours after dosing
Time Frame: Pre-dose (0), and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours post-dose
Population: Not all subjects were available for all bioavailability measurements.
Measure: Number (90% Confidence Interval); unit: Ratio of Adjusted Geometric Means
Groups:
- Regimen B/Regimen A: Single-dose belumosudil 200 mg tablet fed (Regimen B) divided by single-dose belumosudil 200 mg tablet fasted (Regimen A)
Arm/Group | Regimen B/Regimen A | Regimen B/Regimen C
Number analyzed (Participants) | 20 | 20
Ratio of Adjusted Geometric Means
  AUC(0-inf): number analyzed (Participants) | 17 | 17
  AUC(0-inf) | 179.58 [143.16 to 225.26] | 118.43 [97.16 to 144.36]
  AUC(0-last) | 187.92 [154.07 to 229.21] | 117.57 [96.40 to 143.40]
Statistical Analysis 1: Comparison: Regimen B/Regimen A; AUC(0-inf) Null Hypothesis: Ratio of Adjusted Geometric Means = 100%; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, t-test, 2 sided; Ratio of Adjusted Geometric Means (%) = 100, 90% CI 2-sided [80.00 to 125.00]; Intra-subject variability: 34.25%
Statistical Analysis 2: Comparison: Regimen B/Regimen C; AUC(0-inf) Null Hypothesis: Ratio of Adjusted Geometric Means = 100%; Test type: Equivalence — [test comment as in outcome 3, analysis 2]; p = 0.16, t-test, 2 sided; Ratio of Adjusted Geometric Means (%) = 100, 90% CI 2-sided [80.00 to 125.00]; Intra-subject variability;
Statistical Analysis 3: Comparison: Regimen B/Regimen A; AUC(0-last) Null Hypothesis: Ratio of Adjusted Geometric Means = 100%; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; p < 0.001, t-test, 2 sided; Ratio of Adjusted Geometric Means (%) = 100, 90% CI 2-sided [80.00 to 125.00]; Intra-subject variability = 38.16%
Statistical Analysis 4: Comparison: Regimen B/Regimen C; AUC(0-last) Null Hypothesis: Ratio of Adjusted Geometric Means = 100%; Test type: Equivalence — [test comment as in outcome 3, analysis 2]; p = 0.18, t-test, 2 sided; Ratio of Adjusted Geometric Means (%) = 100, 90% CI 2-sided [80.00 to 125.00] — Intra-subject variability = 38.16%; Intra-subject variability = 38.16%

5. Secondary Outcome: Pharmacokinetics: Cmax of Dosing Regimen A (Tablets--Fasting) vs. Dosing Regimen B (Tablets--Fed) vs. Dosing Regimen C (Capsules--Fed) for KD025, KD025m1, and KD025m2 at 48 Hours Post-dose
Description: Maximum concentration (Cmax) of parent drug (KD025), Metabolite 1 (KD025m1), and Metabolite 2 (KD025m2) when administering a single dose of belumosudil 200 mg tablet to subjects who are fasting (Regimen A) compared to administering a single dose of belumosudil 200 mg tablet to subjects who are fed (Regimen B) compared to a single dose of belumosudil 200 mg capsule (two 100-mg capsules) to subjects who are fed (Regimen C) at 48 hours after dosing
Time Frame: Pre-dose (0), and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours post-dose
Population: Based on PK Population: Not all subjects received each regimen.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Regimen C: Single-dose belumosudil 200 mg capsule (two 100-mg capsules) in the fed state
Arm/Group | Regimen A | Regimen B | Regimen C
Number analyzed (Participants) | 23 | 20 | 22
ng/mL
  Cmax: Parent Drug KD025 | 821 (129.5) | 2100 (49.8) | 1750 (38.2)
  Cmax: KD025m1: number analyzed (Participants) | 16 | 20 | 20
  Cmax: KD025m1 | 19.4 (51.6) | 25.8 (42.0) | 20.6 (38.2)
  Cmax: KD025m2: number analyzed (Participants) | 22 | 20 | 22
  Cmax: KD025m2 | 173 (122.6) | 412 (63.0) | 289 (76.5)

6. Secondary Outcome: Pharmacokinetics: AUCs of Regimen A (Tablet--Fasting) vs. Dosing Regimen B (Tablet--Fed) vs. Dosing Regimen C (Capsule--Fed) for KD025, KD025m1, and KD025m2 for Belumosudil 200 mg at 48 Hours Post-dose
Description: Area under concentration curve from zero to last dose (AUC[0-last]) and from zero to infinity (AUC[0-inf]) for parent drug (KD025), Metabolite 1 (KD025m1), and Metabolite 2 (KD025m2) when administering a single dose of belumosudil 200 mg tablet to subjects who are fasting (Regimen A) compared to administering a single dose of belumosudil 200 mg tablet to subjects who are fed (Regimen B) compared to administering a single dose of 200 mg capsule (two 100-mg capsules) to subjects who are fed at 48 hours after dosing
Time Frame: Pre-dose (0), and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours post-dose
Population: Not all subjects in either cohort had all AUC measurements
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (ng*h)/mL
Arm/Group | Regimen A | Regimen B | Regimen C
Number analyzed (Participants) | 23 | 20 | 22
(ng*h)/mL
  AUC(0-last): KD025 | 4520 (121.3) | 9750 (49.3) | 8650 (42.7)
  AUC(0-last): KD025m1: number analyzed (Participants) | 16 | 20 | 20
  AUC(0-last): KD025m1 | 19.8 (150.6) | 45.2 (95.3) | 33.6 (106.9)
  AUC(0-last): KD025m2: number analyzed (Participants) | 22 | 20 | 22
  AUC(0-last): KD025m2 | 550 (133.3) | 1320 (62.6) | 1000 (95.5)
  AUC(0-inf): KD025: number analyzed (Participants) | 14 | 17 | 21
  AUC(0-inf): KD025 | 4910 (146.9) | 10100 (52.9) | 8710 (42.2)
  AUC(0-inf): KD025m1: number analyzed (Participants) | 1 | 1 | 1
  AUC(0-inf): KD025m1 | 153 (0) | 98.7 (0) | 213 (0)
  AUC(0-inf): KD025m2: number analyzed (Participants) | 16 | 17 | 15
  AUC(0-inf): KD025m2 | 691 (76.7) | 1370 (62.6) | 1420 (47.7)

7. Secondary Outcome: Pharmacokinetics: Lambda-z for Regimens A, B, and C for KD025, KD025m1, and KD025m2 at 48 Hours Post-dose
Description: Slope of the regression line passing through the apparent elimination phase in a concentration-time plot (Lambda-z) for Regimen A, Regimen B, and Regimen C for for the parent drug (KD025), Metabolite 1 (KD025m1), and Metabolite 2 (KD025m2) at 48 hours after dosing
Time Frame: Pre-dose (0), and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours post-dose
Population: Not all subjects had PK parameter lambda-z analyzed
Measure: Geometric Mean (Standard Deviation); unit: 1/hour
Arm/Group | Regimen A | Regimen B | Regimen C
Number analyzed (Participants) | 23 | 20 | 22
1/hour
  KD025: number analyzed (Participants) | 14 | 17 | 21
  KD025 | 0.0622 (1.5848) | 0.0993 (1.5293) | 0.0967 (1.4594)
  KD025m1: number analyzed (Participants) | 1 | 1 | 1
  KD025m1 | 0.3618 (0) | 0.3608 (0) | 0.1275 (0)
  KD025m2: number analyzed (Participants) | 16 | 17 | 15
  KD025m2 | 0.4159 (1.5248) | 0.3291 (1.7326) | 0.2523 (1.7385)

8. Secondary Outcome: Pharmacokinetics: t(1/2), MRT(0-last), and MRT(0-inf) for Regimens A, B, and C for KD025, KD025m1, and KD025m2 at 48 Hours Post-dose
Description: Apparent elimination half-life (t[1/2]), mean residence time from zero to last dose (MRT[0-last]), and MRT for zero to infinity (MRT[0-inf]) for Regimen A, Regimen B, and Regimen C for for the parent drug (KD025), Metabolite 1 (KD025m1), and Metabolite 2 (KD025m2) at 48 hours after dosing
Time Frame: Pre-dose (0), and 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours post-dose
Population: Not all subjects had all PK parameters analyzed
Measure: Geometric Mean (Standard Deviation); unit: Hours
Arm/Group | Regimen A | Regimen B | Regimen C
Number analyzed (Participants) | 23 | 20 | 22
Hours
  KD025: t(1/2): number analyzed (Participants) | 14 | 17 | 21
  KD025: t(1/2) | 11.16 (1.58) | 6.98 (1.53) | 7.16 (1.46)
  KD025m1: t(1/2): number analyzed (Participants) | 1 | 1 | 1
  KD025m1: t(1/2) | 1.92 (0) | 1.92 (0) | 5.44 (0)
  KD025m2: t(1/2): number analyzed (Participants) | 16 | 17 | 15
  KD025m2: t(1/2) | 1.67 (1.52) | 2.11 (1.73) | 2.75 (1.74)
  KD025: MRT(0-last) | 7.25 (1.39) | 5.70 (1.27) | 6.21 (1.22)
  KD025m1: MRT(0-last): number analyzed (Participants) | 16 | 20 | 20
  KD025m1: MRT(0-last) | 1.70 (1.61) | 2.45 (1.61) | 2.79 (1.57)
  KD025m2: MRT(0-last): number analyzed (Participants) | 22 | 20 | 22
  KD025m2: MRT(0-last) | 3.03 (1.32) | 3.99 (1.45) | 4.44 (1.34)
  KD025: MRT(0-inf): number analyzed (Participants) | 14 | 17 | 21
  KD025: MRT(0-inf) | 9.35 (1.33) | 6.40 (1.27) | 7.18 (1.24)
  KD025m1: MRT(0-inf): number analyzed (Participants) | 1 | 1 | 1
  KD025m1: MRT(0-inf) | 3.38 (0) | 4.39 (0) | 8.26 (0)
  KD025m2: MRT(0-inf): number analyzed (Participants) | 16 | 17 | 15
  KD025m2: MRT(0-inf) | 3.46 (1.30) | 4.35 (1.46) | 4.86 (1.40)

9. Secondary Outcome: Safety: Number of Subjects With TEAEs and SAEs
Description: Number of subjects with treatment-emergent adverse events (TEAEs), severity and relationship to belumosudil, serious adverse events (SAEs), TEAEs leading to withdrawal from study, and deaths. Treatment-emergent adverse events (TEAEs) are AEs that are not present before the first dose of IMP or that are present before the first dose of IMP but worsen in intensity during exposure to IMP.
  Severity: mild = 1; moderate = 2; severe = 3; life-threatening = 4; and death = 5. Related to belumosudil defined as possibly related, probably related, and related.
Time Frame: Approximately 1 month
Population: All subject who received at least one dose of belumosudil
Measure: Count of Participants; unit: Participants
Groups:
- Regimen A: Single-dose belumosudil 200 mg tablet in the fasted state
  Belumosudil Tablet
- Regimen C: Single-dose belumosudil capsules (administered as two 100-mg capsules) in the fed state
  Belumosudil Capsule
- Overall: Subjects who received Regimen A and/or Regimen B and/or Regimen C
Arm/Group | Regimen A | Regimen B | Regimen C | Overall
Number analyzed (Participants) | 23 | 20 | 22 | 23
Participants
  At least 1 TEAE | 6 | 3 | 5 | 9
  Reporting belumosudil-related TEAEs | 1 | 0 | 0 | 1
  TEAEs Leading to Withdrawal | 3 | 0 | 0 | 3
  Severe TEAEs | 1 | 0 | 0 | 1
  Serious TEAEs | 0 | 0 | 0 | 0
  TEAEs Leading to Death | 0 | 0 | 0 | 0

10. Secondary Outcome: Safety: Total Number of Participants With TEAEs, Related TEAEs, Leading to Withdrawal, Severe, Serious, Leading to Death
Description: Total number of subjects who had treatment-emergent adverse events (TEAEs), TEAEs related to belumosudil, TEAEs leading to withdrawal of subject, severe TEAEs, serious TEAE (SAE), and TEAEs leading to death. Treatment-emergent adverse events (TEAEs) are AEs that are not present before the first dose of IMP or that are present before the first dose of IMP but worsen in intensity during exposure to IMP.
  Severity: mild = 1; moderate = 2; severe = 3; life-threatening = 4; and death = 5. Related to belumosudil defined as possibly related, probably related, and related.
Time Frame: Approximately 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Regimen A | Regimen B | Regimen C | Overall
Number analyzed (Participants) | 23 | 20 | 22 | 23
Participants
  All TEAEs | 7 | 3 | 6 | 16
  TEAEs Related to Belumosudil | 1 | 0 | 0 | 1
  TEAEs Leading to Withdrawal | 3 | 0 | 0 | 3
  Severe TEAEs | 1 | 0 | 0 | 1
  Serious TEAEs (SAE) | 0 | 0 | 0 | 0
  TEAEs Leading to Death | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 1 month
Description: Adverse events were classified into two categories: 1.Pre-dose AEs: AEs recorded at screening or with a start date and time prior to the first does of IMP and either do not continue after or do not worsen in intensity after the first dose of IMP; 2. Treatment-emergent adverse events (TEAEs): AEs that are not present before the first dose of IMP or that are present before the first dose of IMP but worsen in intensity during exposure to IMP.
Arm/Group | Regimen A | Regimen B | Regimen C
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 6/23 | 3/20 | 5/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A (N=23) | Regimen B (N=20) | Regimen C (N=22)
Cervical radiculopathy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Influenza-like illness (General disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 1 | 0 | 0
Transaminase increased (Investigations) | 1 | 0 | 0
Atrioventricular block--2nd degree (Cardiac disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Oropharyngeal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results. The sponsor cannot require changes to the study results in the communication except to remove sponsor's confidential information. Sponsor cannot unilaterally extend the embargo.